CLINICAL TRIAL: NCT02309567
Title: Is There Any Relation Between Serum Anti-p53 Antibody and TLG, MTV and SUV as PET Parameters in Lung Cancer Patients?
Status: Completed | Type: Observational
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Zekiye HASBEK, M.D., Assistant Professor, Cumhuriyet University, School of Medicine, Department of Nuclear Medicine, Cumhuriyet University
Other Study IDs: T-597
Record Dates: First submitted 2014-11-25; First posted 2014-12-05 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Lung Neoplasms; Gene, p53
Keywords: Anti-p53 antibody; PET/CT; Lung Cancer; FDG
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Other: Blood Collection

SUMMARY:
p53 is a tumor suppressor gene which plays an important role in controlling normal cell proliferation regulation that is located on the chromosome 17 (17p13.1). It is the most common goal of genetic alteration in many tumors. Serum p53 protein is presence in normal healthy individuals. However p53 antibody is extremely rare. Mutations in this gene cause an accumulation of non-functional proteins and development of anti-p53 antibodies, which can be detectable in tissues, slouhed cells, blood and other body fluids. Some studies have reported that, p53 mutations are highly common in leukemia, lymphoma, lung, esophagus, stomach, liver, bone, bladder, ovarian, and brain cancers. Lung cancer is the most common cause of cancer-related deaths and the survey is low after the initial diagnosis. Accurate staging is important for determine the choice of treatment and predict prognosis. 18F-FDG PET/BT has important value for initial staging and it is the most advanced imaging technique developed all over the world for determine of the characterization of the metabolic tumor volume. Maksimum Standardized Uptake Value (SUVmax) which was acquired by PET imaging is commonly used in clinical practice as a criterion for malignancy. Due to the development of new software programs recently studies have shown that metabolic tumor volume (MTV) and total lesion glycolysis (TLG) may be useful quantitative parameters for the prognostic evaluation. Viable tumor volume could be estimate with this programs.The purpose of this study was to assess the relation between serum anti-p53 antibody level and quantitative PET parameters as SUVmax, SUVave, MTV and TLG.

ELIGIBILITY:
Inclusion Criteria:

* patients who were referred to our department with the purpose of 18F-FDG PET/CT imaging for staging due to lung cancer diagnosis
* patients who were performed 18F-FDG PET/CT for diagnosis in the cause of the suspected pulmonary nodule/lesion in thorax CT but not detected pathologic FDG accumulation
* In the control group, healthy subjects with no history of cancer and without any complaint

Exclusion Criteria:

* Patients had operated for lung cancer, received prior chemotherapy or radiotherapy for lung cancer, with no definitive histological diagnosis, and a blood glucose level greater than 150 mg/dL

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Lung cancer patients and patients who have suspected pulmonary lesion
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Serum anti-p53 antibody level measurement. | Blood samples for serum anti-p53 antibody will taken before the FDG administration. All serum will immediately frozen and stored. Analysis will performed presumably after 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Cumhuriyet University, School of Medicine, department of Nuclear Medicine, Sivas, Campus, Turkey (Türkiye)